CLINICAL TRIAL: NCT00001640
Title: Genetic Analysis of Parkinson's Disease
Status: Completed | Type: Observational
Sponsor: National Human Genome Research Institute (NHGRI) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 970078; 97-HG-0078
Record Dates: First submitted 1999-11-03; First posted 1999-11-04 (Estimated); Last update posted 2017-07-02 (Actual); Status verified 2009-02-10

CONDITIONS: Parkinson's Disease
Keywords: Parkinson's Disease
MeSH Terms: conditions — Parkinson Disease

SUMMARY:
The purposes of this study are to identify the gene or genes responsible for an inherited form of Parkinson's disease and learn more about how the disease develops.

In Parkinson's disease, a deficiency of a brain chemical called dopamine impairs the function of the part of the brain that controls movement. As a result, patients may have difficulty moving or they may have uncontrolled movements of their hands and fingers. Parkinson's disease usually occurs sporadically, with no known cause. In a few families, however, the disease seems to be inherited through a gene mutation (change). There is a 50-50 chance that a parent with the mutated gene will pass it on to a child. Children who do inherit the abnormal gene may or may not go on to actually develop Parkinson's disease-the relative chance of this happening is not known.

Individuals 18 years of age and older from families in which Parkinson's disease appears to be inherited may be eligible for this study. Participants will have a brief medical examination, provide a personal and family medical history, and have a small blood sample (2 tablespoons) taken for genetic studies. The total time required for the study is about 1 to 2 hours.

Participants are encouraged to meet with a NIH investigator or with a genetics specialist in their local area before testing to talk about the possible implications for themselves and their families of the test results....

DETAILED DESCRIPTION:
Individuals, and where possible multiple family members, from families with inherited Parkinson's disease will be enrolled. We will also be enrolling people with sporadic Parkinson's disease. Known disease genes will be sequenced to look for mutations. In the event that no mutations are detected and there are samples from multiple family members, linkage analysis will be undertaken in an effort to identify a region or regions of the genome harboring defective genes that cause inherited Parkinson's disease. Candidate genes that reside in regions linked to the disease will be sequenced in effort to find mutations responsible for the disease.

Genetic linkage studies will include all available, informative family members, while gene sequence analysis will be performed on affected individuals and spousal controls. In the event that we identify a mutation of clear pathogenicity in one of the known Parkinson's genes, we will contact all participating family members to notify them of the discovery of the gene that causes PD in their family and offer them individual counseling and testing in a CLIA approved lab. To assess any impact caused by the offer and subsequent pursuit of genetic testing we will be administering a questionnaire assessing psychological well-being prior to and following testing.

ELIGIBILITY:
* INCLUSION CRITERIA:

Individuals age 18 or over from families in which an autosomal dominant form of Parkinson's disease is apparently being inherited.

The diagnosis must be supported by accepted clinical criteria: tremor, bradykinesia, and responsiveness to L-DOPA.

Unaffected family members will also be enrolled.

Subjects must give consent.

Parkinson's disease may be associated with dementia.

Decisionally-impaired individuals will be enrolled.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 500
Dates: Start 1997-02-11; Study Completion 2009-02-10

CONTACTS AND LOCATIONS:
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Polymeropoulos MH, Lavedan C, Leroy E, Ide SE, Dehejia A, Dutra A, Pike B, Root H, Rubenstein J, Boyer R, Stenroos ES, Chandrasekharappa S, Athanassiadou A, Papapetropoulos T, Johnson WG, Lazzarini AM, Duvoisin RC, Di Iorio G, Golbe LI, Nussbaum RL. Mutation in the alpha-synuclein gene identified in families with Parkinson's disease. Science. 1997 Jun 27;276(5321):2045-7. doi: 10.1126/science.276.5321.2045. PMID 9197268
- [Background] Polymeropoulos MH, Higgins JJ, Golbe LI, Johnson WG, Ide SE, Di Iorio G, Sanges G, Stenroos ES, Pho LT, Schaffer AA, Lazzarini AM, Nussbaum RL, Duvoisin RC. Mapping of a gene for Parkinson's disease to chromosome 4q21-q23. Science. 1996 Nov 15;274(5290):1197-9. doi: 10.1126/science.274.5290.1197. PMID 8895469
- [Background] Eldridge R, Ince SE. The low concordance rate for Parkinson's disease in twins: a possible explanation. Neurology. 1984 Oct;34(10):1354-6. doi: 10.1212/wnl.34.10.1354. No abstract available. PMID 6541307